CLINICAL TRIAL: NCT00864929
Title: An Epidemiological Study on Antimicrobial Treatment of Nosocomial Infections in Clinical Practice
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca Vietnam
Other Study IDs: NIS-IVN-DUM-2008/1
Record Dates: First submitted 2009-03-18; First posted 2009-03-19 (Estimated); Last update posted 2011-02-16 (Estimated); Status verified 2011-02

CONDITIONS: Nosocomial Infection
Keywords: Non-interventional study; Vietnam; inappropriate treatment; nosocomial infection
MeSH Terms: conditions — Cross Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: Appropriate antimicrobial treatment
- 2: Inappropriate antimicrobial treatment

SUMMARY:
The present study is a retrospective cohort study on patients who suffered a nosocomial infection in major hospitals in Vietnam. Data relating to patient demography include age, gender; medical history; APACHE II score; background conditions, infection details and antimicrobial therapy; and all-caused mortality, time of hospitalization and intensive care. The investigators hypothesis is that antimicrobial treatment inappropriate is highly dependent on incidence of antibiotic resistant pathogens, nonfermentative Gram-negative bacilli and ESBL-producing enterobacteriaceae spp. Variables are demographic characteristics, background conditions, immunosuppressive therapy, antimicrobial susceptibility and inappropriate treatment is explored as possible predictors of mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed as nosocomial infection defined according to criteria established by the US CDC. The diagnosis criteria for ventilator-associated pneumonia are modified from those established by the American College of Chest Physicians.
* Patient received empiric antimicrobial therapy within 24 hour from onset of infection and had antimicrobial susceptibility.

Exclusion Criteria:

* A patient was in part of a controlled clinical trial for the current infection episode.
* Patients with suspected infections by virus or fungus or tuberculosis will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient was diagnosed as nosocomial infection
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
The number and percentage of subjects with nosocomial infection received appropriate antimicrobial treatment | 30 days as from onset of nosocomial infection

SECONDARY OUTCOMES:
The number and percentage of patients with nosocomial infections received de-escalation therapy | 30 days as from onset of nosocomial infection
The number and percentage of hospital mortality, the number of days for hospitalization, intensive care among groups of patients who received appropriate or inappropriate antimicrobial treatments | 30 days as from onset of nosocomial infection
The determinants for inappropriate antimicrobial treatment and mortality. | 30 days as from onset of nosocomial infection

CONTACTS AND LOCATIONS:
Overall Officials: Phan Anh Tuan Nguyen, MD, Study Director — AstraZeneca Vietnam; To Nhu Le, MD, Principal Investigator — National Paediatric Insitute; Viet Hoa Le, Principal Investigator — The 108 Military Central Hospital
Locations (2):
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City